CLINICAL TRIAL: NCT03701646
Title: Comparing Non-invasive Cardiac Output Measurements by the ClearSight Hemodynamic Monitoring System to Thermodilution Measurements in Pediatric Patients Undergoing Cardiac Catheterization.
Brief Title: ClearSight Validation in Pediatrics
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1146179
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Shock; Hypotension and Shock
MeSH Terms: conditions — Shock; Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- arterial line: Pediatric patients admitted to the ICU with a medically indicated arterial line.
  Interventions: Device: Measurement by Clearsight device
- cardiac output: Pediatric patients requiring cardiac output measurement by thermodilution through cardiac catheterization.
  Interventions: Device: Measurement by Clearsight device

INTERVENTIONS:
Device: Measurement by Clearsight device — Clearsight Device is used to obtain non-invasive measurements to be correlated to standard invasive measurements.

SUMMARY:
Specific aim 1: The specific aim of this study is to compare cardiac output measurements as well as cardiac index, and stroke volume obtained via thermodilution during a cardiac catheterization with data obtained by the ClearSight cardiac output monitoring system. Specific aim 2: To compare arterial blood pressure measurements obtained by arterial line with arterial waveform measurements obtained by the ClearSight System. The hypothesis is: Cardiac output measurements or arterial blood pressure measurements taken non-invasively with the ClearSight system in pediatric patients who are either undergoing cardiac catheterization or have an arterial line will correlate with cardiac output measurements taken by pulmonary artery catheter thermodilution or arterial pressures measured by an arterial line.

DETAILED DESCRIPTION:
Specific aim number one: To compare cardiac output measurements obtained from the Clear Sight cardiac output monitor with measurements obtained with thermodilution in the cardiac catheterization laboratory. Significance: Currently, based on the Surviving Sepsis guidelines, fluid administration is supposed to be guided by measurements of fluid responsiveness. Currently, there are very few ways to obtain measurements of fluid responsiveness, such as cardiac output, stroke volume, and systemic vascular resistance non-invasively. The invasive methods are no longer used in pediatrics, as the risk of placing these invasive catheters is felt to outweigh the benefit of using the data provided by the invasive cardiac output monitoring systems. Although the Clear Sight cardiac output monitoring system has been validated in adults to measure cardiac output non-invasively, this technology has not been evaluated in pediatrics. If the Clear Sight monitoring system is shown to be accurate in pediatrics, it would safely provide data that could be lifesaving to a pediatric patient in shock.

Specific aim number two: To compare the accuracy of the Clear Sight cardiac output monitor in obtaining continuous blood pressure measurements non-invasively. Significance: Currently, the only reliable method to continuously monitor blood pressure in critically ill patients is with an invasive intra-arterial catheter. Placing this catheter carries risks with it, including risk of infection as well as risk of intra-arterial thrombus which can lead to limb ischemia. The Clear Sight cardiac output monitor has the technology to obtain continuous blood pressure measurements non-invasively, although this technology has never been validated in pediatric patients. Therefore, specific aim 1 is to determine if this technology can reliably be used in pediatric patients. If it can, this would provide a method to obtain continuous blood pressure measurements without the risk of an invasive catheter.

Hypothesis: Cardiac output and arterial blood pressure measurements taken non-invasively with the ClearSight system in will correlate with cardiac output measurements taken by pulmonary artery catheter thermodilution and arterial blood pressure measurements taken by arterial line. This hypothesis is based on personal communications with the developers of this device.

ELIGIBILITY:
Arm 1) Cardiac output measurements Patients will be selected as potential study participants from the patients undergoing cardiac catheterization in the Nemours Cardiac Center for medically indicated reasons.

Patients selected should meet the following criteria:

* Age 17 years old or younger
* Receiving a cardiac catheterization, including cardiac output measurement, for clinical purposes, as determined by their cardiologist
* Hemodynamically stable with a scheduled non-emergent catheterization

Patients will be excluded from this study if:

* have digits too small to effectively fit into the smallest ClearSight finger probe
* Are hemodynamically unstable

Arm 2) Arterial blood pressure measurements

Patients will be selected as potential study participants from the patients admitted to the pediatric intensive care unit and now requiring an arterial line for medically indicated reasons.

Patients selected should meet the following criteria:

- Age 17 years old or younger

Patients will be excluded from this study if:

- Have digits too small to effectively fit into the smallest ClearSight finger probe

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients admitted to the ICU requiring an arterial line, or patients undergoing cardiac output measurements by cardiac catheterization by thermodilution.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Measurement of non-invasive cardiac output or continuous blood pressure correlated to invasive measurements. | 11/2/2017 - 6/1/2019
  Comparison of measurements obtained by the ClearSight device compared to the invasive measurements will be used to evaluate whether the ClearSight device has any validity in pediatrics.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours A.I. duPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No